CLINICAL TRIAL: NCT06926244
Title: RESistance of IgA Nephropathy to Conventional and Newly-approved Therapies: an Observational, Real-life Study (RESIGAN)
Acronym: RESIGAN
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP 240615
Record Dates: First submitted 2025-03-03; First posted 2025-04-13 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: IgA Nephropathy (IgAN)
Keywords: IgAN; Primary Glomerulonephritis; Mesangial IgA Deposits
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
IgA nephropathy (IgAN) is the most common primary glomerulonephritis worldwide, characterized by glomerular mesangial IgA deposits, often with IgG and C3. Despite its prevalence, the pathophysiology of IgAN is poorly understood. The prognosis varies significantly, from benign hematuria to rapidly progressive glomerulonephritis, potentially leading to end-stage renal disease within months. The MEST-C classification enhances prognosis characterization and informs integrated scoring systems; however, while useful for assessing overall prognosis, these scores do not reliably predict treatment responses and are unvalidated for IgA vasculitis nephritis. Given the disease's heterogeneity, treatment options for IgAN, with or without vasculitis, are controversial. Nephroprotective strategies that lower intraglomerular pressure through RAS blockade are essential in managing IgAN. Steroids are considered for rapidly progressive cases, yet their effectiveness in persistent proteinuria despite optimized nephroprotection is debated. Other immunosuppressive therapies, such as B cell targeting and complement inhibition, are under investigation. Recently developed nephroprotective strategies, including SGLT2 inhibitors and endothelin-1 receptor antagonists, may significantly influence future therapeutic approaches. Although available in many European countries, their real-world effectiveness has not been evaluated. Identifying factors linked to persistent proteinuria and renal dysfunction despite optimized nephroprotection is a critical unmet need. We hypothesize that innovative nephroprotective strategies will reduce the risk of persistent proteinuria and renal dysfunction in an IgAN cohort.

DETAILED DESCRIPTION:
IgA Nephropathy (IgAN) is the most prevalent primary glomerulonephritis globally, diagnosed by detecting mesangial IgA deposits in the kidneys, often accompanied by IgG and C3. The disease's pathophysiology remains unclear despite its commonality. Prognosis can vary widely, from benign hematuria to rapidly progressive forms leading to end-stage renal disease within months. The MEST-C classification provides histological prognostic factors that enhance prognosis assessment and facilitate the development of integrated scoring systems. However, these scores are limited in predicting treatment responses and lack validation for IgA vasculitis nephritis.

Given the disease's heterogeneity, treatment strategies for IgAN are contentious. Nephroprotective approaches focusing on reducing intraglomerular pressure through RAS blockade play a significant role in management. Steroids are suggested for rapidly progressive disease, but their effectiveness in persistent proteinuria, despite optimized nephroprotection, is debated. Other treatments, including B cell-targeting therapies and complement inhibition, are under investigation. Recent advances in nephroprotection, such as SGLT2 inhibitors and endothelin-1 receptor antagonists, could significantly reshape future therapeutic strategies. While these treatments are widely available in Europe, their real-world effectiveness remains to be evaluated. Identifying factors linked to persistent proteinuria and renal dysfunction despite optimized strategies is a pressing unmet need.

This study hypothesizes that new nephroprotective strategies will influence the risk of persistent proteinuria and renal dysfunction in a real-life cohort of IgAN patients.

Primary Objective: To identify clinical, biological, and histological risk factors for persistent proteinuria and renal dysfunction in IgAN patients.

Secondary Objectives include:

Identifying risk factors for steroid therapy response. Evaluating responses to nephroprotective therapies, including SGLT2 inhibition. Analyzing responses to immunosuppressive therapies at various time points post-diagnosis.

Assessing risk factors for persistent proteinuria and renal dysfunction in patients with related conditions or IgA vasculitis.

Identifying risk factors for adverse events following nephroprotection or immunosuppressive therapies.

Describing treatment trajectories since IgAN diagnosis. Validating the International IgA Nephropathy prediction tool. Developing a cohort of IgAN patients will facilitate reliable epidemiological data collection and allow for the evaluation of responses to contemporary treatments, identifying patients with treatment resistance in real-life scenarios. This identification is critical for establishing early, efficient therapeutic strategies for IgAN patients at risk of progression.

Study Design: A prospective and retrospective observational cohort study.

Inclusion Criteria:

Adult patients aged ≥ 18 years. Renal biopsy after 2017 confirming IgA deposits for IgAN diagnosis (index date).

Informed consent from patients who do not object to data use. Non-inclusion Criteria: None.

Cohort Details:

Retrospective Cohort: Expected 600 patients, inclusion from 01/01/2017 to study start date.

Prospective Cohort: 200 participants over 2 years, followed for 2 years, totaling 4 years of research.

For retrospective data collection, information notes will be mailed to patients, allowing data use after one month without opposition. Prospective patients will receive study information during clinic visits, with data used if there is no objection. Data will be extracted from medical records, including clinical, histological, and laboratory results, collected by clinical research assistants or investigators. Patient Health Information (PHI) will be stored securely, with only month and year of birth recorded for privacy.

Analysis: For primary outcomes, univariable analysis will utilize logistic regression to explore the association of risk factors with outcomes. A multivariable model may be developed based on expert knowledge and univariable results. The model's performance will be assessed via the area under the curve (AUC) and R², with bootstrap validation to evaluate for overfitting.

Total Research Duration: 4 years, with a recruitment period of 2 years and a follow-up period of 2 years. The retrospective data will cover at least 2 years post-IgAN diagnosis, potentially extending up to 12 years based on the biopsy date (from 2017).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient: age ≥ 18 years
* Renal biopsy performed after 2017 showing IgA deposits leading to the diagnosis of IgAN (the date of diagnosis being the index date)
* Informed patient and who does not object to the use of his data

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 800 patients is expected:
  * Retrospective cohort: 600 patients to be expected : Renal biopsy showing IgA deposits leading to the diagnosis of IgAN performed from 2017 to date of start of the study
  * Prospective cohort: 200 participants : Renal biopsy showing IgA deposits leading to the diagnosis of IgAN performed from the date of start of the study : 1 to 2patients with new diagnosis/ site/month
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with persistent proteinuria (>1 g/g) and/or renal dysfunction (>20% eGFR decline) at twelve months from diagnosis. | month 12 from diagnosis
  Persistent proteinuria is defined as protein/creatinine ratio >1 g/g; renal dysfunction is defined as a loss of >20% eGFR (Estimated Glomerular Filtration Rate) as compared to eGFR measured at baseline.

SECONDARY OUTCOMES:
Proportion of patients with persistent proteinuria (>1 g/g) and/or renal dysfunction (>20% eGFR decline) at 6 months from diagnosis | month 6 from diagnosis
  Persistent proteinuria is defined as protein/creatinine ratio >1 g/g; renal dysfunction is defined as a loss of >20% eGFR (Estimated Glomerular Filtration Rate) as compared to eGFR measured at baseline.
Proportion of patients with persistent proteinuria (>1 g/g) and/or renal dysfunction (>20% eGFR decline) at twenty-four months from diagnosis. | month 24 from diagnosis
  Persistent proteinuria is defined as protein/creatinine ratio >1 g/g; renal dysfunction is defined as a loss of >20% eGFR as compared to eGFR measured at baseline.
Proportion of patients with persistent proteinuria (>1 g/g) and/or renal dysfunction (>20% eGFR decline) at the end of follow-up. | At the end of follow-up, that is at least 2 years from inclusion
  Persistent proteinuria is defined as protein/creatinine ratio >1 g/g; renal dysfunction is defined as a loss of >20% eGFR as compared to eGFR measured at baseline.
Proportion of patients experiencing a Major Adverse Renal Event (MARE) by month 12, defined as the initiation of dialysis, receipt of a kidney transplant, or onset of renal failure | month 12 from diagnosis
  Major Adverse Renal Events will be defined as the occurrence of any of the following events at the time of assessment:
  * Renal failure, defined as a loss of more than 40% in eGFR as compared to the initial eGFR or eGFR <15 ml/min/1.73m2
  * Dialysis
  * Transplantation
Proportion of patients experiencing a Major Adverse Renal Event (MARE) by month 6, defined as the initiation of dialysis, receipt of a kidney transplant, or onset of renal failure | month 6 from diagnosis
  Major Adverse Renal Events will be defined as the occurrence of any of the following events at the time of assessment:
  * Renal failure, defined as a loss of more than 40% in eGFR as compared to the initial eGFR or eGFR <15 ml/min/1.73m2
  * Dialysis
  * Transplantation
Proportion of patients with absence of response to steroids therapy defined as persistent proteinuria or renal dysfunction at the end of steroids treatment | At the end of steroids treatment, that is on average at 6 months from inclusion
  Persistent proteinuria is defined as protein/creatinine ratio >1 g/g; renal dysfunction is defined as a loss of >20% eGFR as compared to eGFR measured at baseline.
Proportion of patients with severe hyperkalemia (>6mM/l) evaluated at each visit | Baseline, Month 3, Month 6, Month 12, Month 24, and then each year until the end of follow-up
  Severe hyperkalemia defined as hyperkalemia > 6mM/l
Proportion of patients with severe acute renal failure (KDIGO stage 3) at each visit until the end of follow-up | Baseline, Month 3, Month 6, Month 12, Month 24, and then each year until the end of follow-up
  Acute renal failure diagnosis reaching criteria of the stage 3 of the KDIGO classification:
  * Serum creatinine 3.0 times baseline
  * Serum creatinine ≥ 4.0 mg/dl
  * Initiation of renal replacement therapy
Proportion of patients with 50% decline in eGFR or end-stage kidney disease at any time during follow-up | Baseline, Month 3, Month 6, Month 12, Month 24, and then each year until the end of follow-up
  * Loss of more than 50% in eGFR as compared to the initial eGFR
  * End-stage kidney disease, defined as eGFR <15 ml/min/1.73m2

CONTACTS AND LOCATIONS:
Locations (1):
- Nephrology department, Hospital Pitié - Salpêtrière (ASSISTANCE PUBLIQUE HOPITAUX DE PARIS AP-HP), Paris, France

IPD SHARING:
Plan to Share IPD: Undecided